CLINICAL TRIAL: NCT07381556
Title: The Effectiveness of Cyclosporine Versus Methotrexate in the Treatment of Pediatric Alopecia Areata in Routine Clinical Care: a Patient Preference Trial
Brief Title: Cyclosporine Or Methotrexate for Pediatric Alopecia Areata: Routine Clinical Care Effectiveness Study
Acronym: COMPARE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Rick Waalboer-Spuij, MD, PhD, Deputy Head of Department of Dermatology, MD, PhD., Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2025-0562
Record Dates: First submitted 2026-01-07; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata(AA); Alopecia Areata (AA); Alopecia Totalis/Universalis; Alopecia Universalis (AU); Alopecia Totalis (AT); Alopecia Areata (& Ophiasis)
Keywords: Pediatric; Alopecia areata; systemic treatment alopecia areata
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — Methotrexate; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (MTX) (Active Comparator): Methotrexate is administered orally or intramusculairly and dosed 10-15mg/m2, 1 times a week, with folate suppletion 24 hours after MTX intkae
  Interventions: Drug: Methotrexate
- Cyclosporine (Cyclo) (Active Comparator): Cyclosporine is given orally, dosed 3-5mg/kg/day and divided in to two doses/ day
  Interventions: Drug: Cyclosporin (CSA)

INTERVENTIONS:
Drug: Methotrexate — MTX is given at a dose of 10-15mg/m2 per week, orally or subcutaneously. Additionally, folate supplementation is administered concurrently as part of standard care, with folate 5-10 mg/week administered 24 hours after MTX intake.
  Arms: Methotrexate (MTX)
Drug: Cyclosporin (CSA) — CSA is given orally (tablet or liquid form) and dosed 3-5mg/kg/day, divided into two doses a day
  Arms: Cyclosporine (Cyclo)

SUMMARY:
Rationale: Since the introduction of Janus kinase (JAK) inhibitors, there has been a significant advancement in the treatment of pediatric alopecia areata. Eligibility for this treatment, in the Netherlands, requires prior failure of systemic therapies such as cyclosporin or methotrexate. However, the choice between methotrexate and cyclosporin as first-line systemic treatment is not supported by robust comparative studies.

Therefore, the investigators conduct a patient preference trial with a long-term follow-up provided in the Pediatric Systemic Alopecia Areata Registry (STA2R-Pediatric). This study will evaluate the effectiveness of Cyclosporin (CsA) and Methotrexate (MTX) in children and adolescents with moderate-to-severe AA.

Objective(s): To investigate the effectiveness of CsA and MTX in the treatment of children and adolescents with alopecia areata in routine clinical care.

Study type: This is a prospective, patient preference clinical trial with a duration up to 36 weeks in accordance with the routine clinical care guidelines.

Study population: This study will include children and adolescents (2-17 years old) diagnosed with AA who start first-line systemic treatment.

Methods: Patients and their parents will choose between CsA and MTX treatment as in routine clinical care, receiving follow-up in accordance with standard clinical practices. The participants will not be randomized. The primary endpoint is the measurement of the Severity of Alopecia Tool (SALT) at 9-months with a secondary endpoint at 24 weeks. SALT scores will be measured by a blinded assessor. The (Children) - Dermatology Life Quality Index ((C)-DLQI) questionnaire will be conducted at each visit (0, 3, 6, 9 months), allowing evaluation of the impact on patients' quality of life.

DETAILED DESCRIPTION:
Rationale: Alopecia areata (AA) is a dermatological disorder characterized by non-scarring hair loss, significantly affecting the quality of life of patients. While some patients experience spontaneous hair regrowth or respond well to localized treatments, patients with moderate-to-severe AA represent a subgroup that requires systemic therapies for effective management. If the disease is severe and systemic treatment is desired, cyclosporine or methotrexate is initiated. Currently, the clinical management of moderate-to-severe AA is primarily based on expert opinions. There is a lack of research on systemic treatments for moderate-to-severe AA, comprising only a small number of randomized controlled trials and observational studies. There is a clear absence of long-term, prospective, and comparative data on these systemic therapies. Most conventional systemic treatments for AA are prescribed off-label, underlining the importance of gaining a more comprehensive understanding of their effectiveness and safety.

Since the introduction of Janus kinase (JAK) inhibitors, there has been a significant advancement in the treatment of pediatric alopecia areata. As of 2024, Ritlecitinib-a selective JAK3 inhibitor-has been approved for reimbursement in adolescents aged 12 years and older with severe disease (defined as SALT50 or greater). Eligibility for this treatment requires prior failure of systemic therapies such as cyclosporin or methotrexate. However, the choice between methotrexate and cyclosporin as first-line systemic treatment is not supported by robust comparative studies and is largely based on expert opinion, resulting in considerable (inter)national variation in clinical practice.

Therefore, the investigators conduct a patient preference trial with a long-term follow-up provided in the Pediatric Systemic Alopecia Areata Registry (STA2R-Pediatric). This study will evaluate the effectiveness of Cyclosporin (CsA) and Methotrexate (MTX) in children and adolescents with moderate-to-severe AA. Aiming to provide valuable insights into the effectiveness, safety, and long-term outcomes of these therapies. By collecting and analyzing such data, this study endeavors to contribute to evidence-based clinical management, ultimately improving care for children and adolescents with AA.

Objective(s): To investigate the effectiveness of CsA and MTX in the treatment of children and adolescents with alopecia areata in routine clinical care.

Study type: This is a prospective, patient preference clinical trial with a duration up to 36 weeks in accordance with the routine clinical care guidelines after which patients will be followed in the STA2R-Pediatric (PANAMA-ID 11347).

Study population: This study will include children and adolescents (2-17 years old) diagnosed with AA who start first-line systemic treatment.

Methods: Patients and their parents will choose between CsA and MTX treatment as in routine clinical care, receiving follow-up in accordance with standard clinical practices. They will not be randomized. The primary endpoint is the measurement of the Severity of Alopecia Tool (SALT) at 9-months, providing a quantitative assessment of the disease's activity and response to the selected treatment. SALT scores will be measured by a blinded assessor. The (Children) - Dermatology Life Quality Index ((C)-DLQI) questionnaire will be conducted at each visit (0, 3, 6, 9 months), allowing evaluation of the impact on patients' quality of life.

Burden and risks: Participants in this study will receive treatment according to standard clinical practice protocols. The only addition to their routine care will be one questionnaire at each visit, that takes no more than 5 minutes to complete. The investigators consider this to be a negligible risk.

Recruitment and consent: Eligible patients will be identified at the dermatology outpatient clinic. During a routine visit to the outpatient clinic, the dermatologist will explain the study to the patient and the patient will be asked whether they would be willing to participate in the study. Patients will have the opportunity to ask any questions to clarify their understanding and concerns about the study. The Patient Information Form, Informed Consent Form, and instructions on how to proceed if they are interested in taking part or finding out more about the study will be given to the patient and their parents. During this visit the physician involved in the study will inform the patients and answer all the questions, Informed Consent can be obtained during the same visit. The Informed Consent will be completed and signed by the patient, their parents, and the physician. For patients under 12 years of age, consent will be signed by the parents only.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age 2-17 years
* Clinical diagnosis of AA by a certified dermatologist
* Willingness of participant (in case 12-17 years) and parents to provide informed consent for participation in the study.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Inability to adhere to the study protocol, including medication intake, clinic visits, and questionnaire completion.
* Patients who are ineligible for the CsA arm (due to contraindications), are automatically included in the MTX arm.
* Contra-indications CsA:

Impaired kidney function. Poorly controlled hypertension Active infections. Presence of a malignancy. Nephrotic syndrome combined with poorly controlled hypertension, infection or malignancy.

Kidney disorders, except in cases of nephrotic syndrome with mild to moderate renal impairment.

* Patients who are ineligible for the MTX arm (due to contraindications), are automatically included in the CsA arm.
* Contraindications MTX:

Conception (both male and female) and lactation Severe kidney or liver dysfunction (fibrosis, cirrhosis) or alcohol abuse Bone marrow hypoplasia, immunodeficiency Anemia, leukopenia, or thrombocytopenia Poor nutritional status (low albumin) Hypersensitivity or allergy to MTX Lung toxicity due to MTX or significant reduction in lung function.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
SALT 36 weeks | 36 weeks
  To compare SALT* (delta-SALT and SALT<20) between baseline and 36 weeks of treatment between the CsA and MTX group.
  * The Severity of Alopecia Tool (SALT) score is a standardized, numerical measure (0-100) used by dermatologists to quantify scalp hair loss in patients with alopecia areata. A score of 0 indicates no hair loss, while 100 indicates total scalp hair loss.

SECONDARY OUTCOMES:
SALT 24 weeks | 24 weeks
  To compare SALT* (delta- SALT and SALT<20) between CsA and MTX at 24 weeks.
  * The Severity of Alopecia Tool (SALT) score is a standardized, numerical measure (0-100) used by dermatologists to quantify scalp hair loss in patients with alopecia areata. A score of 0 indicates no hair loss, while 100 indicates total scalp hair loss.
Quality of life (DLQI) | 24, 36 weeks
  To compare the quality of life c-DLQI* or DLQI* between CsA and MTX at 0, 12, 24, 36 weeks.
  *DLQI = Dermatology Life Quality Index, measures impact of skin diseases on a patient's life. The score ranges from 0 (no impact) to 30 (extreme impact).
Adverse events | 0, 12, 24, 36 weeks
  To compare side effects in CSA and MTX group.
Discontinuation of therapy | 0, 12, 24, 36 weeks
  To compare the proportion of patients who discontinued therapy in CSA and MTX group.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided